CLINICAL TRIAL: NCT03425435
Title: Quality of Care of Oncological Patients With Home Parenteral Nutrition
Brief Title: Quality of Care of Oncological Patients With HPN
Acronym: VHPE-S
Status: Terminated | Type: Observational
Why Stopped: preterm stop due to low recruitment numbers during and still ongoing pandemic
Sponsor: Fresenius Kabi (Industry)
Responsible Party: Sponsor
Other Study IDs: HPNM-001-CNI
Record Dates: First submitted 2018-02-01; First posted 2018-02-07 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Tumors and Home Parenteral Nutrition
MeSH Terms: conditions — Neoplasms | interventions — Quality of Life; Health Services Research

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: QoL and developed questionnaires for healthcare research — Questionnaires

SUMMARY:
Medical care for patients with home parenteral nutrition (HPN) is challenging. Among other aspects, the transition from the inpatient to the outpatient setting (discharge management), the organization of HPN at home or in a care facility (care management), the expertise required to care for patients with HPN and consistent compliance with standards are key to the quality of care for patients requiring HPN.

Hospital patients on parenteral nutrition (PN) to be continued at home are often discharged at very short notice. A good interlocking of all players is required to collect and distribute the relevant information, to secure proper training for those involved and to have all utilities and equipment at hand when the patient arrives.

This study collects nutritional and clinical parameters (including patient-reported parameters) along the continuum of care of HPN patients to evaluate the impact of the quality of care of HPN patients on their quality of life.

DETAILED DESCRIPTION:
The HPN management will be evaluated by using a self-developed patient and a standardized quality of life questionnaire.

Patients will be recruited at the participating hospital by their treating physician before discharge and will continue their study participation after discharge.

The documentation period for the individual patients will be 3 months.

The questions of the patient´s questionnaire cover areas of interest like: satisfaction with discharge management, nutrition, satisfaction with HPN.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with an initial prescription for HPN during the current hospital stay
* Planned PN must at least contain the macronutrients glucose and amino acids.
* Solid, malignant tumor
* Anticipated duration of the HPN is at least 28 days
* Age ≥18 years
* Full legal capacity or legal guardian available
* Fluent in German language
* Able to read and write in German language
* Signed patient informed consent form
* Indication for PN

Exclusion Criteria:

* Contraindication for PN
* ECOG performance status >3
* Pregnant and breast-feeding women
* Concurrent participation in another clinical study that requires deviations from the hospital's routine PN, nutrition and/or nursing procedures

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with solid tumors with indication for home parenteral nutrition.
Sampling Method: Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2022-01-14 (Actual)

PRIMARY OUTCOMES:
Patient´s questionnaire | Outcome measures obtained 1, 4 and 12 weeks after discharge from hospital
  Mean changes in total scores of QoL-questionnaire from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Schneider, Dr. med., Principal Investigator — Hannover Medical School, Germany
Locations (1):
- Medizinische Hochschule Hannover, Hanover, Germany

REFERENCES:
- [Derived] Schneider A, Baur C, Zopf Y, Torok HP, Sina C, Prinz C, Monnich H, Madisch A, Maluck-Scholecke S, Rotzer I, Seipt C, Gotte A, Beer J, Jager E. Quality of care of oncological patients with home parenteral nutrition. Support Care Cancer. 2024 Nov 29;32(12):834. doi: 10.1007/s00520-024-09011-2. PMID 39612012